CLINICAL TRIAL: NCT05399498
Title: An Open Label Study of Single-Dose Psilocybin for Major Depressive Disorder With Co-occurring Borderline Personality Disorder
Brief Title: Psilocybin in Co-occuring Major Depressive Disorder and Borderline Personality Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0272
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Borderline Personality Disorder; Major Depressive Disorder
Keywords: BPD; MDD; Psilocybin
MeSH Terms: conditions — Borderline Personality Disorder; Depressive Disorder, Major | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Open-label treatment study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Psilocybin (Experimental): Single 25 mg capsule oral dose of psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin 25mg capsule

SUMMARY:
The primary objective of the study is to evaluate the safety and efficacy of psilocybin in adults with major depressive disorder (MDD) and borderline personality disorder (BPD).

DETAILED DESCRIPTION:
The primary objective of the proposed study is to evaluate the safety and efficacy of psilocybin in adults with major depressive disorder (MDD) and borderline personality disorder (BPD). Ten subjects with MDD and BPD will receive a single 25 mg oral dose of psilocybin. The hypothesis to be tested is that psilocybin will result significant reduction in symptoms of both MDD and BPD after 1 week and sustained for 4 weeks compared to baseline (improvement in symptoms will be indicated by lower scores on established outcome measures of MDD and BPD symptoms that have been used in prior studies).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Diagnosed with current major depressive disorder
* Montgomery-Asberg Depression Rating Scale (MADRS) score of > 20
* Diagnosed with borderline personality disorder
* Borderline Personality Disorder Symptom Assessment Scale (BPD-SAS) score of > 20
* Ability to understand and sign the consent form

Exclusion Criteria:

* Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
* Illegal substance use based on urine toxicology screening (except cannabis use)
* Current or past history of bipolar I disorder, schizophrenia, or schizoaffective disorder
* Active substance use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline to Week 5
  One of the co-primary outcome measures will be the change from baseline using the Montgomery-Asberg Depression Rating Scale (MADRS). The MADRS is a 10-item, clinician-administered scale that assesses depression symptoms during the last seven days. Each item is rated on a scale from 0 to 6, with 0 being "normal/not present" and 6 being "extreme."
Borderline Personality Disorder Symptom Assessment Scale (BPD-SAS) | Baseline to Week 5
  One of the co-primary outcome measures will be the change from baseline using the Borderline Personality Disorder Symptom Assessment Scale (BPD-SAS). The BPD-SAS covers a two-week time frame and each of the nine criteria, each representing symptoms of BPD, for BPD is rated on a five-point anchored rating scale of 0-4, with 0 representing no symptoms and 4 representing extreme symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity scale (CGI-S) | Baseline to Week 5
  A clinician administered, single item scale measuring global severity of psychiatric illness. The scale itself assesses overall disorder severity on a scale from 1 to 7 with 1 being "not at all" and 7 being "among the most severe cases"
Clinical Global Impression - Improvement scale (CGI-I) | Week 2 to Week 5
  A clinician administered, single item scale measuring overall improvement of global severity of psychiatric illness. The scale itself assesses overall disorder improvement on a scale from 1 to 7 with 1 being "Very much improved" and 7 being "Very much worse"

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunderson J: Borderline Personality Disorder, 2nd ed. Washington, DC, American Psychiatric Press, 2000
- [Background] Nakao K, Gunderson JG, Phillips KA, Tanaka N: Functional impairment in personality disorders. J Pers Disord 1992; 6:24-31
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] Blum N, St John D, Pfohl B, Stuart S, McCormick B, Allen J, Arndt S, Black DW. Systems Training for Emotional Predictability and Problem Solving (STEPPS) for outpatients with borderline personality disorder: a randomized controlled trial and 1-year follow-up. Am J Psychiatry. 2008 Apr;165(4):468-78. doi: 10.1176/appi.ajp.2007.07071079. Epub 2008 Feb 15. PMID 18281407
- [Background] McMain SF, Guimond T, Streiner DL, Cardish RJ, Links PS. Dialectical behavior therapy compared with general psychiatric management for borderline personality disorder: clinical outcomes and functioning over a 2-year follow-up. Am J Psychiatry. 2012 Jun;169(6):650-61. doi: 10.1176/appi.ajp.2012.11091416. PMID 22581157
- [Background] Lieb K, Vollm B, Rucker G, Timmer A, Stoffers JM. Pharmacotherapy for borderline personality disorder: Cochrane systematic review of randomised trials. Br J Psychiatry. 2010 Jan;196(1):4-12. doi: 10.1192/bjp.bp.108.062984. PMID 20044651
- [Background] Nickel MK, Muehlbacher M, Nickel C, Kettler C, Pedrosa Gil F, Bachler E, Buschmann W, Rother N, Fartacek R, Egger C, Anvar J, Rother WK, Loew TH, Kaplan P. Aripiprazole in the treatment of patients with borderline personality disorder: a double-blind, placebo-controlled study. Am J Psychiatry. 2006 May;163(5):833-8. doi: 10.1176/ajp.2006.163.5.833. PMID 16648324
- [Background] Schulz SC, Zanarini MC, Bateman A, Bohus M, Detke HC, Trzaskoma Q, Tanaka Y, Lin D, Deberdt W, Corya S. Olanzapine for the treatment of borderline personality disorder: variable dose 12-week randomised double-blind placebo-controlled study. Br J Psychiatry. 2008 Dec;193(6):485-92. doi: 10.1192/bjp.bp.107.037903. PMID 19043153
- [Background] Zanarini MC, Schulz SC, Detke HC, Tanaka Y, Zhao F, Lin D, Deberdt W, Kryzhanovskaya L, Corya S. A dose comparison of olanzapine for the treatment of borderline personality disorder: a 12-week randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2011 Oct;72(10):1353-62. doi: 10.4088/JCP.08m04138yel. PMID 21535995
- [Background] Pascual JC, Soler J, Puigdemont D, Perez-Egea R, Tiana T, Alvarez E, Perez V. Ziprasidone in the treatment of borderline personality disorder: a double-blind, placebo-controlled, randomized study. J Clin Psychiatry. 2008 Apr;69(4):603-8. doi: 10.4088/jcp.v69n0412. PMID 18251623
- [Background] Zanarini MC, Vujanovic AA, Parachini EA, Boulanger JL, Frankenburg FR, Hennen J. Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD): a continuous measure of DSM-IV borderline psychopathology. J Pers Disord. 2003 Jun;17(3):233-42. doi: 10.1521/pedi.17.3.233.22147. PMID 12839102